CLINICAL TRIAL: NCT02930538
Title: Can Postoperative Outcomes be Predicted From Asking OSA Screening Questions Pre-operatively?
Status: Withdrawn | Type: Observational
Why Stopped: PI left the institution
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Vidya Raman, Clinical Associate Professor of Anesthesiology, Nationwide Children's Hospital
Other Study IDs: IRB16-00491
Record Dates: First submitted 2016-09-15; First posted 2016-10-12 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children undergoing surgery: Children ages 3-18 undergoing a surgical procedure at Nationwide Children's Hosp.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Completing a survey on RedCap

SUMMARY:
The proposed research will determine whether a 6-item screening questionnaire previously shown to correlate with moderate or severe OSA is useful for predicting postoperative outcomes in children undergoing surgery under general anesthesia.

DETAILED DESCRIPTION:
The survey will be administered preoperatively in the ENT clinic or the preoperative surgical unit. The following data will also be recorded: patient demographics (age, gender, BMI), surgical procedure, length of procedure and anesthetic, and smoking exposure. Based on differences in postoperative outcomes (e.g., supplemental oxygen requirement in the PACU) observed in the derivation cohort for the 6-item questionnaire, the study will enroll 1,000 patients to attain sufficient power for evaluating the 6-item questionnaire in the overall cohort and in demographically or clinically defined subgroups.

ELIGIBILITY:
Inclusion Criteria:

* The study will include all who are presenting for surgery to the main operating room, ambulatory surgical center or procedure center at Nationwide Children's Hospital.

Exclusion Criteria:

* Emergency surgery and any caregiver or patient refusal.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children having surgery at Nationwide Children's Hosp (NCH).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Liters of Oxygen | 1 hr post-op
  The patient's oxygen requirement while in the PACU.

SECONDARY OUTCOMES:
Narcotic usage in mg | 1 hr post-op
  The patient's opiod requirement while in the PACU.
PACU length of stay | 1-2 hr post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided